CLINICAL TRIAL: NCT07370311
Title: A Culturally Adapted Decision Aid Intervention to Support Chinese American Dementia Caregivers in Feeding-Related Decisions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007171
Record Dates: First submitted 2026-01-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dementia Caregivers; End of Life Decision Making; Advanced Dementia
Keywords: Chinese Americans; feeding options; decision aid; decision coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participation Group (No Intervention): 1. Receive usual care (including information from healthcare providers)
  2. Receive electrical version of decision aid after all of the data collection
- Intervention/Treatment Group (Experimental): 1. Receive both the electronic and paper version of CMCFODA
  2. Receive an individualized decision coaching within two weeks
  Interventions: Other: Chinese version of Making Choices Feeding Options for Patients with Dementia Decision Aid

INTERVENTIONS:
Other: Chinese version of Making Choices Feeding Options for Patients with Dementia Decision Aid — Participants in the treatment group will receive the CMCFODA via zoom meeting or another secure video conferencing platform and an individualized decision coaching.
  Arms: Intervention/Treatment Group

SUMMARY:
Family caregivers of people with dementia have to decide between tube feeding and hand feeding when persistent eating problems arise. This decision can be difficult for Chinese American dementia caregivers, due to the interplay of culture, potential absence of a patient's advance directive, poor understanding of dementia, and lack of knowledge on the risks and benefits of tube feeding. In this polit study, the principal investigator examines whether a culturally adapted decision aid intervention regarding feeding options named "Chinese version of Making Choices Feeding Options for Patients with Dementia Decision Aid" (CMCFODA) will improve Chinese American caregivers' decision-making about feeding options in patients with moderate or advanced dementia. The proposed study advances the field by providing critical evidence to inform the development and implementation of culturally adapted decision support interventions in end-of-life dementia care.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Self-identify as Chinese
* Providing caregiving or involvement in end-of-life care decision-making for older Chinese adults with: a) moderate or advanced dementia, b) feeding difficulties, and c) poor oral intake, eating/swallowing problems, or weight loss

Exclusion Criteria:

* Dementia patients are a) receiving tube feeding, b) enrolled in hospice care, or 3) have a documented preference against a feeding tube

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Decision conflict | Baseline; One-Month Follow-Up; Three-Month Follow-Up
  SURE test for decisional conflict (0-4)
Knowledge of feeding options and dementia | Baseline; One-Month Follow-Up; Three-Month Follow-Up
  Questions to assess knowledge about feeding options and dementia
Expectations of tube feeding | Baseline; One-Month Follow-Up; Three-Month Follow-Up
  Questions about understanding differing expectations regarding feeding tube use

SECONDARY OUTCOMES:
Frequency of communication with other family members and healthcare providers | Baseline; One-Month Follow-Up; Three-Month Follow-Up
  Questions to understand caregiver involvement, support, and information flow
Preference of feeding option | Baseline; One-Month Follow-Up; Three-Month Follow-Up
  Careful hand feeding, tube feeding, or unsure
Preparation for decision-making scale (treatment group only) | One-Month Follow-Up; Three-Month Follow-Up
  Questions to assess the effect of the intervention by preparing for feeding option decision-making
The Feasibility of the CMCFODA study as measured by recruitment rates and the proportion of participants that decline participation. | Enrolment
  The feasibility of the CMCFODA study will be measured by the proportion of eligible participants who decline to participate among those who were screened into the study.
The Feasibility of the CMCFODA study as measured by participant retention, as indicated by the number of participants lost to follow-up. | Enrollment to 3-month Follow-Up
  Participant retention, as an aspect of feasibility, will be measured by the recorded number of participants number lost to follow-up.
Acceptability of the decision aid and decision coaching (only for the treatment group) | One month follow-up
  We will use developed questions to measure the acceptability of this intervention

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the CMCFODA study will be shared only after the investigators have published findings addressing the study's specific aims. Intellectual property and data generated under this project will be managed in accordance with University of Texas at Austin and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance. Following publication of the investigators' primary findings, access to the study databases and associated decision aid intervention tools will be made available for educational, research, and non-profit purposes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: These data will be shared after the investigators have published the study's specific aims. Requests to access the code for this study will be reviewed by the investigative team and granted once feasibility, acceptability, and preliminary efficacy have been evaluated and the findings have been published.
Access Criteria: Individuals who wish to access the data must agree to: (1) use the data solely for research purposes; (2) not attempt to identify any individual participant; (3) securely store the data using appropriate safeguards, such as password-protected servers and files; and (4) return and/or destroy the data upon completion of analyses.